CLINICAL TRIAL: NCT06826105
Title: Effect of Low Dose Pancrelipase With an Oral Nutritional Supplement to Improve Nutrient Bioavailability in Patients at Increased Risk of Malnutrition
Brief Title: Pancrelipase With Nutritional Supplement in Patients at Risk of Malnutrition (EFFORT-ENZO)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipp Schuetz (Other)
Responsible Party: Sponsor-Investigator, Philipp Schuetz, Prof. MD, Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-02519; ka24Schuetz
Record Dates: First submitted 2025-02-03; First posted 2025-02-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Malnutrition
Keywords: Pancrelipase; Oral nutritional supplements
MeSH Terms: conditions — Malnutrition | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pancrelipase (Experimental): two capsules each containing 15000 USP units of lipase
  Interventions: Drug: Zenpep
- Placebo (Placebo Comparator): two capsules each containing placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zenpep — two capsules (each containing 15000 USP units of lipase) together with nutritional supplements
  Other Names: Pancrelipase
  Arms: Pancrelipase
Drug: Placebo — two capsules (containing placebo) together with nutritional supplements
  Other Names: lactose monohydrate
  Arms: Placebo

SUMMARY:
This study investigates if pancreatic enzymes in combination with oral nutritional supplement can improve nutrient bioavailability in older people with malnutrition or at risk of malnutrition.

DETAILED DESCRIPTION:
This study investigates whether adding digestive pancreatic enzymes to oral nutritional supplements (ONS) can improve nutrient absorption in older adults at risk of malnutrition. While ONS are commonly recommended, their effectiveness is often limited due to age-related declines in exocrine pancreatic function, leading to reduced enzyme secretion. Studies indicate that pancreatic lipase levels decline with age, potentially impairing nutrient digestion and absorption.

The study proposes using pancrelipase (Zenpep®), an FDA-approved pancreatic enzyme replacement therapy, to enhance nutrient bioavailability. The randomized, placebo-controlled trial will assess whether pancrelipase improves postprandial levels of amino acids, fatty acids, and glucose in hospitalized patients at nutritional risk.

The study aims to determine if pancreatic enzyme supplementation can enhance nutrient absorption and provide a novel strategy for managing malnutrition in older adults without diagnosed exocrine pancreatic insufficiency (EPI). If successful, this approach could improve clinical outcomes, reduce healthcare costs, and enhance quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Male or female 70 years of age or older
* Hospitalized at site
* Nutrition Risk Screening 2002 (NRS-2002) ≥ 3
* eGFR ≥ 30 mL/min/1.73 m2 (EPI-CKD) based on medical history (no older than 6 months)
* Ability to eat orally

Exclusion Criteria:

* Patients with acute cardiovascular event ≤ 2 days
* Patients with terminal conditions
* Patients diagnosed with pancreatic exocrine insufficiency (EPI) treated with pancreatic enzyme replacement therapy (PERT)
* Patients having a planned transplant or new-onset dialysis in the next 6 months.
* Patients having a colectomy, resection of the small intestine or cholecystectomy
* Known hypersensitivity to any of the substances or excipients of the ONS or the medicinal product

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incremental area under the curve of total branched-chained amino acid concentration | From oral nutritional supplements (ONS) consumption over 3 hours postprandial, specifically in 5 time points (T0 ONS consumption and after 30, 60, 120 and 180 minutes)
  Evaluation of the incremental area under the curve (iAUC) of total branched-chain amino acid (BCAA) concentration in blood, including leucine (μmol/L), isoleucine (μmol/L), and valine (μmol/L). The iAUC represents the time-dependent changes in BCAA levels and is used to assess metabolic responses.

SECONDARY OUTCOMES:
Incremental area under the curve of essential amino acids (EAAs) | From ONS consumption over 3 hours postprandial, specifically in 5 time points (T0 ONS consumption and after 30, 60, 120 and 180 minutes)
  Evaluation of the incremental area under the curve (iAUC) of essential amino acids (EAAs) in plasma, expressed in micromoles per liter (μmol/L). The iAUC reflects the time-dependent changes in EAAs concentrations and is used to assess metabolic responses.
Incremental area under the curve of total amino acids | From ONS consumption over 3 hours postprandial, specifically in 5 time points (T0 ONS consumption and after 30, 60, 120 and 180 minutes)
  Evaluation of the incremental area under the curve (iAUC) of total amino acids in plasma, expressed in micromoles per liter (μmol/L). The iAUC reflects the time-dependent changes in total amino acid concentrations and is used to assess metabolic responses.
Incremental area under the curve of free fatty acids | From ONS consumption over 3 hours postprandial, specifically in 5 time points (T0 ONS consumption and after 30, 60, 120 and 180 minutes)
  Evaluation of the incremental area under the curve (iAUC) of free fatty acids in plasma, expressed in micromoles per liter (μmol/L). The iAUC reflects the time-dependent changes in free fatty acid concentrations and is used to assess metabolic responses.
Incremental area under the curve of triglycerides | From ONS consumption over 3 hours postprandial, specifically in 5 time points (T0 ONS consumption and after 30, 60, 120 and 180 minutes)
  Evaluation of the incremental area under the curve (iAUC) of triglycerides in plasma, expressed in millimoles per liter (mmol/L). The iAUC reflects the time-dependent changes in triglycerides concentrations and is used to assess metabolic responses.
Water load satiety test (WLST) | From ONS consumption over 3 hours postprandial, specifically in 5 time points (T0 ONS consumption and after 30, 60, 120 and 180 minutes)
  Values of a modified water load satiety test (WLST), a questionnaire of 5 sub-scores on a scale of 1-100. We will report both the sum of the scores and the 5 individual sub scales will be reported. Participant rate pre-and postprandial intensity of symptoms for fullness, hunger, abdominal discomfort, bloating, and nausea on a 0-100 mm visual analogue scale where 0 is none, and 100 is severe
Exploratory subgroup analysis | After study completion, within 1 year
  Exploratory subgroup analyses to test their effect on the primary outcome (incremental area under the curve (AUC) of total branched-chained amino acid concentration in the blood) will be performed. These will be assessed using a t-test on the differences between pancrelipase and placebo for each patient. Groups are based on the subgroup including median age [years], malnutrition risk [Nutritional Risk Screening 2002 total score], median weight [kg], sex [male/female], prior history of gastrointestinal side effects [yes/no], median fecal elastase [μg/g]
Incremental area under the curve of glucose | From ONS consumption over 3 hours postprandial, specifically in 5 time points (T0 ONS consumption and after 30, 60, 120 and 180 minutes)
  Evaluation of the incremental area under the curve (iAUC) of glucose in plasma, expressed in millimoles per liter (mmol/L). The iAUC reflects the time-dependent changes in glucose concentrations and is used to assess metabolic responses.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Schuetz, Prof. MD, Principal Investigator — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Switzerland